CLINICAL TRIAL: NCT04901403
Title: Earned Income Tax Credit Access Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Katie Maguire-Jack, Associate Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00190754
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: The Study is Intended to Increase Take-up of EITC
MeSH Terms: interventions — Educational Status; House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education intervention (Other): Parents in the treatment group will receive information about Earned Income Tax Credit, including how to sign up for free. They will also receive help with budgeting and finances from their home visitor.
  Interventions: Other: Education; Other: Home visiting
- Control group (Other): Control group families will receive home visiting services as usual.
  Interventions: Other: Home visiting

INTERVENTIONS:
Other: Education — Parents will be provided with information about Earned Income Tax Credits and budgeting
  Arms: Education intervention
Other: Home visiting — Parents as Teachers home visiting program

SUMMARY:
The EITC Access Study an intervention study provided to families in 7 counties in Michigan.The intervention involves appending a concentrated benefits advocacy intervention onto an existing home visiting program. There are 5 treatment counties and 2 control counties that will survey families in the home visiting program to compare the relative benefits of the added benefits advocacy intervention on the outcomes of parent mental health, intimate partner violence, economic hardship, earned income tax credit take-up, and child maltreatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age, has a child in their home

Exclusion Criteria:

* Does not speak or read English, Spanish, Burmese, or Arabic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Earned Income Tax Credit receipt | Within 2 years of receiving the intervention
  Self-report

SECONDARY OUTCOMES:
Child maltreatment behaviors | Within 2 years of receiving the intervention
  Self-report on the Brief Child Abuse Potential Inventory. 34 Yes/No questions. E.g. "A child needs very strict rules."
Intimate partner violence | Within 2 years of receiving the intervention
  Self-report from Women's Experiences of Battering Scale. 10 items relating to how they would describe their life with their partner. Scale ranges from Strongly agree to strongly disagree. E.g. 1. He makes me feel unsafe even in my own home.
Depression | Within 2 years of receiving the intervention
  Self-report from the Center for Epidemiologic Studies Depression Scale (CES-D). 20 questions on a scale from "rarely" to "most or all of the time" relating to things experienced within the past week. E.g. "I was bothered by things that usually don't bother me."
Anxiety | Within 2 years of receiving the intervention
  Self-report from the General Anxiety Disorder (GAD-7). 7 questions relating to feelings experienced over the past 2 weeks, with response options ranging from "not at all" to "nearly every day." E.g. "Not being able to stop or control worrying."
Economic hardship | Within 2 years of receiving the intervention
  Self-report on 11 yes or no items indicating whether individual hardships were experienced in the past year. E.g. "Was there anyone in your household who needed to see a doctor or go to the hospital but could not go because of the cost?"

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Calhoun Intermediate School District, Battle Creek, Michigan
  - SOS Community Services, Belleville, Michigan
  - Sanilac Intermediate School District, Croswell, Michigan
  - Keweenaw Family Resource Center, Houghton, Michigan
  - Catholic Charities Diocese of Kalamazoo, Kalamazoo, Michigan
  - St Clair RESA, Marysville, Michigan
  - Kalamazoo KRESA, Portage, Michigan

IPD SHARING:
Plan to Share IPD: No
Only aggregate information will be shared with other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT04901403/ICF_000.pdf